CLINICAL TRIAL: NCT00812110
Title: Influenza Vaccination for Parents and Other Caregivers in the Pediatric Medical Home
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 081105
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza prevention
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Influenzae vaccine — 0.5 mL Deltoid Intramuscular Injection X 1
  Other Names: Fluzone

SUMMARY:
We hypothesize that when offered influenza vaccine at little or no cost, in a setting where the value of the vaccine is connected to one's high risk child, vaccination rates for parents will approach 90-95%, similar to rates obtained in the Neonatal Intensive Care Unit environment.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregiver adults who accompany at-risk children to a Pediatric Care outpatient clinic appointment. High risk children are defined as those 0 to 5 years of age, or who have any of the following diagnoses:

  * Sickle cell disease
  * Asthma
  * Cystic fibrosis
  * Chronic renal disease
  * Congenital heart disease
  * Cancer
  * Any immunodeficiency

Exclusion Criteria:

* Caregivers of children residing in group homes
* Persons whose children do not meet the Center for Disease Control (CDC) definition of high-risk
* Persons who have had allergic reactions to influenza vaccination or any other vaccination in the past
* Persons who are allergic to eggs or egg products
* Persons who are allergic to thimerosol
* Previous diagnosis of Guillain-Barré syndrome (GBS)
* Persons who are moderately to severely ill at the time the vaccination is to be given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C White, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the 2008-2009 influenza season, 474 caregivers were approached. 292 agreed to participate,and had not received influenza vaccine.
Groups:
- Caregivers: Caregivers of children at high risk, per CDC definitions, of complications of influenza.
Period: Overall Study
Arm/Group | Caregivers
Started | 292
Completed | 292
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Caregivers
Number analyzed (Participants) | 292
Age Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 171
  White | 100
  More than one race | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 292

OUTCOME MEASURES:

1. Secondary Outcome: Background Rate of Influenza Vaccination in the Parents/Caregivers of High Risk Pediatric Patients in a Low Income Population?
Description: Number of participants who received influenza vaccine the prior year.
Time Frame: 16 months
Measure: Number; unit: participants
Groups:
- Caregivers: Caregivers of children at risk for complications of influenza
Arm/Group | Caregivers
Number analyzed (Participants) | 292
participants | 69

2. Primary Outcome: Number of Participants Who Received Influenza Vaccine.
Description: Caregivers identified for participation were offered influenza vaccine. This describes the number who accepted vaccination
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Caregivers
Number analyzed (Participants) | 292
participants | 250

ADVERSE EVENTS:
Arm/Group | Caregivers
Serious Adverse Events (participants affected / at risk) | 0/292
Other Adverse Events (participants affected / at risk) | 0/292

LIMITATIONS AND CAVEATS:
Exclusively urban,lower socioeconomic status population limits external generalizability. Study was uncontrolled; historical controls were referenced instead. Baseline vaccination rates were self-reported. Possible bias in at-risk determination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes